CLINICAL TRIAL: NCT00618761
Title: Insulin Secretory Capacity in Insulin-independent Pancreas-Kidney Recipients Compared to Non-Diabetic Kidney Recipients, Insulin Independent Recipients of Beta-cell Grafts and Healthy Controls.
Brief Title: Insulin Secretory Capacity in Insulin-independent Pancreas-Kidney Recipients Compared to Controls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Pieter Gillard, Prof Dr, University Hospital, Gasthuisberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: clamp01; JDRF 4/2005/1327
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2008-01

CONDITIONS: Kidney Transplantation; Pancreas Transplantation
Keywords: glucose clamp; beta-cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): kidney-pancreas recipients
  Interventions: Other: hyperglycemic clamp test
- 2 (Active Comparator): kidney recipients
  Interventions: Other: hyperglycemic clamp test
- 3 (Active Comparator): healthy controls
  Interventions: Other: hyperglycemic clamp test
- 4 (Active Comparator): beta-cell recipients
  Interventions: Other: hyperglycemic clamp test

INTERVENTIONS:
Other: hyperglycemic clamp test — hyperglycemic clamp test

SUMMARY:
The purpose of this study is to compare functional beta-cell mass using the hyperglycaemic clamp test in insulin-independent pancreas-kidney recipients with that in non-diabetic kidney recipients and normal controls as well as with the partially previously reported data in beta-cell recipients.

ELIGIBILITY:
Inclusion Criteria:

* kidney pancreas recipients
* kidney recipients
* healthy volunteers
* beta-cell recipients
* immunosuppression with MMF-Tacrolimus
* 1-4 years after transplantation

Exclusion Criteria:

* high doses of steroids
* insulin dependent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
insulin secretion during clamp test | time 0

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Mathieu, M.D., PhD, Principal Investigator — UZ-Gasthuisberg, Department of Endocrinology
Locations (1):
- Department of Endocrinology, Leuven, UZ-Gasthuisberg, Leuven, Belgium